CLINICAL TRIAL: NCT04215731
Title: Neoadjuvant mFOLFOXIRI Plus Bevacizumab Versus Induction FOLFOX Followed by Concomitant Chemoradiotherapy in Patients With High-Risk Locally Advanced Rectal Cancer: Multicenter Randomized Phase III Trial
Brief Title: Neoadjuvant mFOLFOXIRI Plus Bevacizumab in Patients With High-Risk Locally Advanced Rectal Cancer
Acronym: FOBEAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yanhong Deng (Other)
Responsible Party: Sponsor-Investigator, Yanhong Deng, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIHSYSU-17
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy; Bevacizumab; Oxaliplatin; Irinotecan; Fluorouracil; Leucovorin; Chemoradiotherapy; Surgical Procedures, Operative; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOXIRI Plus Bevacizumab (Experimental): Patients will receive neoadjuvant mFOLFOXIRI plus bevacizumab once every two weeks for 4 cycles and the same mFOLFOXIRI for 2 cycles. After completing all 6 cycles chemotherapy, the patient will have an MRI scan to examine the tumor. If MRI restaging is ycT4a/b, or MRF involved, the patient will receive concomitant chemoradiotherapy (preoperative radiotherapy consisted of 50 Gy in 25 fractions, and concurrent with capecitabine at a fixed dose of 825 mg/m2 twice daily on days 1 to 5 for 5 weeks). If MRI restaging is ycT0-3 and MRF negative, then the patient will proceed directly to surgery.
  Interventions: Drug: Neoadjuvant chemotherapy with mFOLFOXIRI plus bevacizumab; Procedure: Restaging; Procedure: Surgery; Radiation: Chemoradiotherapy (only when patients with MRF involved or ycT4a/b by restaging)
- Induction FOLFOX Followed by Concomitant Chemoradiotherapy (Active Comparator): Patients will receive induction FOLFOX chemotherapy for 4 cycles and followed by concomitant chemoradiotherapy (preoperative radiotherapy consisted of 50 Gy in 25 fractions, and concurrent with capecitabine at a fixed dose of 825 mg/m2 twice daily on days 1 to 5 for 5 weeks), then the patient will proceed to surgery.
  Interventions: Radiation: Concomitant Chemoradiotherapy; Procedure: Surgery; Drug: Induction chemotherpay with FOLFOX

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy with mFOLFOXIRI plus bevacizumab — Bevacizumab (5 mg/kg on day 1) plus mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 150 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) for 4 cycles and mFOLFOXIRI (oxaliplatin 85 mg/m2, irinotecan 150 mg/m2, and folinic acid 400 mg/m2 followed by 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) for 2 cycles
  Other Names: Oxaliplatin; Irinotecan; 5-Fluorouracil; Leucovorin; Bevacizumab
  Arms: mFOLFOXIRI Plus Bevacizumab
Procedure: Restaging — Restaging by pelvic magnetic resonance imaging (MRI)
  Arms: mFOLFOXIRI Plus Bevacizumab
Radiation: Concomitant Chemoradiotherapy — Concomitant chemoradiotherapy (preoperative radiotherapy consisted of 50 Gy in 25 fractions, and concurrent with capecitabine at a fixed dose of 825 mg/m2 twice daily on days 1 to 5 for 5 weeks)
  Arms: Induction FOLFOX Followed by Concomitant Chemoradiotherapy
Procedure: Surgery — Radical surgery (TME or more extended surgery)
Radiation: Chemoradiotherapy (only when patients with MRF involved or ycT4a/b by restaging) — Chemoradiotherapy (preoperative radiotherapy consisted of 50 Gy in 25 fractions, and concurrent with capecitabine at a fixed dose of 825 mg/m2 twice daily on days 1 to 5 for 5 weeks)
  Arms: mFOLFOXIRI Plus Bevacizumab
Drug: Induction chemotherpay with FOLFOX — mFOLFOX6 (oxaliplatin 85 mg/m2, and folinic acid 400 mg/m2 followed by bolus 5-fluorouracil 400 mg/m2 and 5-fluorouracil 2400mg/m2 as a 46-hour continuous infusion on day 1) for 4 cycles
  Other Names: Oxaliplatin; 5-Fluorouracil; Leucovorin
  Arms: Induction FOLFOX Followed by Concomitant Chemoradiotherapy

SUMMARY:
Multimodality treatment that comprises preoperative fluoropyrimidine with concurrent radiotherapy followed by total mesorectal excision (TME) surgery and adjuvant fluoropyrimidine-based chemotherapy is recommended as a standard treatment of patients with stage II/III rectal cancer. However, the main target of radiotherapy is local control but no improvement in disease-free survival (DFS) or overall survival (OS) has been shown with this treatment strategy, which leaves approximately 30% of patients in whom distant metastases will develop. Moreover, the short- and long-term adverse effects of radiotherapy such as chronic pain, faecal incontinence and urogenital/anal dysfunction are associated with poor quality of life.

Neadajuvant chemotherpay (NACT) alone has been proposed instead of preoperative chemoradiotherapy (CRT) with the aim of elimination of potential micrometastasis as early as possible while avoiding the adverse effects of radiotherapy, without jeopardizing local control.

Evidence from the UK CR07 trial suggests that, without RT, a local recurrence rate of 5% (27/543) can be achieved if a complete mesorectal excision is carried out with a negative CRM. A small single-center phase II pilot trial treated patients with stage II or III rectal cancer with induction FOLFOX/bevacizumab chemotherapy followed by CRT only in those with stable or progressive disease and resection in all patients. All 32 of the participants had an R0 resection, and the 4-year DFS was 84%. Another phase II trial, which included 60 patients with stage II/III rectal cancer, assessed the R0 resection rate after FOLFOX plus either bevacizumab or cetuximab. An R0 resection was achieved in 98.3% of the participants, and the pathologic complete response rate was 16.7%. The phase III FOWARC trial, compared neoadjuvant therapy with and without radiation and found that perioperative mFOLFOX6 alone led to a similar downstaging rate as fluorouracil-radiotherapy, and no significant difference in outcomes was found between mFOLFOX6 without radiotherapy and 5-FU- radiotherapy.

On the basis of the results of these trials, The investigators hypothesized that radiotherapy could be selectively omitted for patients who respond to NACT alone. The results of TRIBE showed that FOLFOXIRI plus bevacizumab yield a high objective response rate (ORR) (65%), early tumor shrinkage (ETS) (62.7%) and depth of response (DoR) (43.4%) in patients with metastatic colorectal cancer.

The investigators were motivated to investigate this triplet-drugs chemotherpay plus bevacizumab both by the possibility of avoiding the toxicities of radiation without compromising local control, and the possibility that earlier introduction of intensive systemic therapy might achieve rapid tumor shrinkage, and improve distant control.

The investigators conducted this phase III trial to compare neoadjuvant mFOLFOXIRI plus bevacizumab with selective radiotherapy with induction FOLFOX followed by concomitant chemoradiotherapy in patients with high-risk locally advanced rectal cancer.

DETAILED DESCRIPTION:
This trial is a two-arm, multicenter, open labelled, prospective, randomized phase III studies. Eligible patients with high-risk locally advanced rectal cancer patients (cT3 with any MRF involved, any cT4a/b or lateral node positive) will be randomly assigned, in a 1:1 ratio, to receive either neoadjuvant mFOLFOXIRI plus bevacizumab with selective radiotherapy or induction FOLFOX followed by concomitant chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Histological or cytological documentation of adenocarcinoma of the rectal (<12 cm from the anal verge).
3. Determined preoperatively by pelvic MRI: high risk locally advanced (cT3 with any MRF involved, any cT4a/b, or lateral node positive).
4. Male or female subjects > 18 years < 70 of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. CT or MRI scans (done within 30 days of registration) of the chest, abdomen and pelvis all without clear evidence of distant metastatic (M1) disease.
7. Non complicated primary tumor (complete obstruction, perforation, bleeding).
8. No previous any systemic anticancer therapy for colon cancer disease.
9. Adequate bone marrow, hepatic and renal function as assessed by the following laboratory requirements conducted within 7 days of starting study treatment:

Exclusion Criteria:

1. Previous or concurrent cancer that is distinct in primary site or histology from colon cancer within 5 years prior to randomization.
2. Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment.
3. Heart failure grade III/IV (NYHA-classification).
4. Unresolved toxicity higher than CTCAE v.4.0 Grade 1 attributed to any prior therapy/procedure.
5. Subjects with known allergy to the study drugs or to any of its excipients.
6. Current or recent (within 4 weeks prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
7. Breast- feeding or pregnant women
8. Lack of effective contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | up to 3 years
  Defined as the time from randomization to relapse or death, whichever occurred first.

SECONDARY OUTCOMES:
R0 resection rate | up to 3 years
  R0 resection defined as complete tumor resection with all margins being negative.
Pathologic complete response | up to 3 years
Overall survival (OS) | up to 5 years
  Defined as the time from randomization to death from any cause.
Toxicity assessed using the NCI common toxicity criteria, version 4.0. | up to 5 years
  The grade of toxicity will be assessed using the NCI common toxicity criteria, version 5.0.
Postoperative morbidity | up to 5 years
local recurrence rate | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No